CLINICAL TRIAL: NCT00006372
Title: Phase I Trial of Combination Pegylated Liposomal Doxorubicin (Doxil), Vinorelbine, and Gemcitabine
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Beth A. Overmoyer, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1Y99; P30CA043703 (NIH); CWRU-1Y99; NCI-G00-1859
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Patients receive gemcitabine IV over 30 minutes on days 1 and 8. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.
Drug: pegylated liposomal doxorubicin hydrochloride — Patients receive doxorubicin HCl liposome IV over 1-2.5 hours on day 1. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.
Drug: vinorelbine ditartrate — Patients receive vinorelbine IV over 6-10 minutes on days 1 and 15. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pharmacokinetic profile of gemcitabine, doxorubicin HCl liposome, and vinorelbine in patients with advanced solid tumors.
* Determine the maximum tolerated dose of this regimen in these patients.
* Determine the toxicity profile of this regimen in these patients.

OUTLINE: This is a dose escalation study.

Patients receive doxorubicin HCl liposome IV over 1-2.5 hours on day 1, gemcitabine IV over 30 minutes on days 1 and 8, and vinorelbine IV over 6-10 minutes on days 1 and 15. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome, gemcitabine, and vinorelbine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

Patients are followed every 3 months for up to 1 year.

PROJECTED ACCRUAL: Approximately 9-24 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor not amenable to curative surgery, radiotherapy, or chemotherapy
* No brain metastases or primary brain tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,500/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin no greater than 1.2 mg/dL
* AST and/or ALT less than 2.5 times upper limit of normal (ULN)
* PT no greater than ULN (anticoagulant independent)

Renal:

* Creatinine no greater than 1.5 mg/dL AND/OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease
* LVEF at least 45% by MUGA or echocardiogram

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow or peripheral blood stem cell transplantation following high dose chemotherapy
* At least 3 weeks since prior biologic therapy for cancer and recovered
* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy:

* See Disease Characteristics
* See Biologic therapy
* No more than 1 prior chemotherapy regimen
* No prior vinca alkaloids
* Prior anthracycline allowed if total dose no greater than 300 mg/m2
* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or carmustine) and recovered

Endocrine therapy:

* At least 3 weeks since prior endocrine therapy for cancer and recovered

Radiotherapy:

* See Disease Characteristics
* No more than 1 prior radiotherapy regimen
* At least 4 weeks since prior large field radiotherapy
* At least 3 weeks since prior radiotherapy for cancer and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2000-02; Primary Completion 2003-04 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth A. Overmoyer, MD, FACP, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States